CLINICAL TRIAL: NCT05413213
Title: Efficiency of an Ambulatory Rehabilitation Program in Patients With Shoulder Degenerative Rupture of the Rotator Cuff Tendons
Brief Title: Ambulatory Rehabilitation Program in Patients With Degenerative Rupture of the Rotator Cuff Tendons of the Shoulder
Acronym: ERARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: APHP200070
Record Dates: First submitted 2022-05-02; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain; rotator cuff tendons; Ambulatory rehabilitation
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Experimental group: Ambulatory rehabilitation program based on mobilizations and muscular solicitations (muscle strengthening and dynamic humeral recentering), supervised by a physiotherapist, consisting of 15 individual sessions of 30 minutes each, spread over 8 weeks, according to a standardized program .
  Control group: Ambulatoryrehabilitation program, consisting of ultrasound physiotherapy, supervised by a physiotherapist, consisting of 15 individual sessions of 30 minutes each, spread over 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The experimental plan is that of therapeutic research. This is a multicenter, prospective, comparative, randomized patient study in 2 parallel arms (ratio 1: 1) in single blind, providing for 134 participants.
  They can provide an unbiased evaluation of the effect of this intervention, randomisation having the effect of eliminating any influence of the patient or the doctor on the allocation of the intervention and therefore of not guiding the selection of patients according to the intervention they will receive. Conducting a double-blind trial would be impossible here. The patient and the physiotherapist will be aware of the treatment arm to which the patient belongs. However, the evaluator (who is not the therapist) will not know the treatment arm and the patient will not know the hypothesis tested (effectiveness of the rehabilitation received by the experimental group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Ambulatory rehabilitation program based on mobilization and muscular solicitation
  Interventions: Procedure: Ambulatory rehabilitation program
- Control Group (Active Comparator): Ambulatory rehabilitation program using ultrasound physiotherapy
  Interventions: Procedure: Ambulatory rehabilitation program

INTERVENTIONS:
Procedure: Ambulatory rehabilitation program — Experimental group: Ambulatory rehabilitation program based on mobilization and muscular solicitation.

SUMMARY:
The main objective of the research is to study the effectiveness of an ambulatory rehabilitation program based on mobilization and muscular solicitation, during painful shoulders by full-thickness degenerative rupture of the tendons of the rotator cuff. , with the algo-functional state, ie pain and activity limitation, as judgment criteria, at 3 months.

DETAILED DESCRIPTION:
Our hypothesis is that rehabilitation based on mobilization and muscular solicitation is effective in painful shoulder due to degenerative rupture of the tendons of the rotator cuff; that it reduces pain, functional limitation and the need for surgery.

Research Excluding health products:

Experimental group: Ambulatory rehabilitation program based on mobilization and muscular solicitation

Control group: Ambulatory rehabilitation program using of ultrasound physiotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 55 years old,
2. Painful shoulder for at least 1 month,
3. Shoulder treated with at least one cortisone infiltration one month or more before inclusion,
4. Pain ≥ 40/100 on visual analog scale,
5. Pain reproduced by at least one clinical test of rotator cuff tendons or subacromial impingement (Jobe, Patte, Neer, Yocum test, Hawkins),
6. Full-thickness tear of at least one tendon of the rotator cuff attested by imaging,
7. Affiliation to social security

Exclusion Criteria:

1. Passive glenohumeral mobility of the shoulder limited,
2. Calcifying tendinopathy on standard radiography,
3. Glenohumeral arthropathy;
4. Painful acromioclavicular arthropathy;
5. History of shoulder fracture;
6. Neurogenic pain or neurogenic motor deficit of the upper limb;
7. Cortisone infiltration of the shoulder in the month preceding inclusion;
8. Operated shoulder;
9. Systemic pathologies including inflammatory rheumatism or neoplastic pathology;
10. Patient participating in another experimental research;
11. Patient under legal protection (curators or guardianship)
12. Patient deprived of liberty by a judicial or administrative decision
13. Pregnant or breastfeeding woman

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain | At 3 month follow-up
  algo-functional scorec SPADI, measured with Visual Analog Score
Shoulder disability | At 3 month follow-up
  algo-functional score SPADI, measured with Visual Analog Score

SECONDARY OUTCOMES:
Shoulder active mobility | 3, 6, 12 months
  Pain subscore of the SPADI scale
  Abduction strength by dynamometer, Activity limitation by the function subscore of the SPADI scale , Life quality Overall improvement perceived by the patient by the 5-point Likert scale, at 3 months, 6 months and 1 year; The total algo-functional score of the SPADI scale at 6 months and 1 year; The use of non-surgical care, Assessed by drug consumption, the number of cortisone infiltrations, The number of non-protocol rehabilitation sessions and the number of consultations outside the scope of the study; The use of surgery for degenerative rupture of the tendons of the rotator cuff by the number of surgical interventions and the Type of surgery performed in this indication during follow-up, The time off work by the number of days

CONTACTS AND LOCATIONS:
Overall Officials: BEAUDREUIL Johann, Pr, Study Chair — Lariboisière Hospital -physical medicine and rehabilitation department